CLINICAL TRIAL: NCT05124626
Title: Chest Wall Motility in Pectus Excavatum Patients Before and After MIRPE Performed With One or Two Metallic Bars: a Comparative Study
Brief Title: Evaluation of Chest Wall Motility After MIRPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital Alemão Oswaldo Cruz (Other); Traumec Tecnologia e Implantes Ortopedicos Ltda (Unknown)
Responsible Party: Principal Investigator, Miguel L. Tedde, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29724420.1.0000.0068
Record Dates: First submitted 2021-10-05; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Funnel Chest
Keywords: Funnel chest; Quality of life; Video-assisted thoracic surgery; Prostheses and implants.
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One bar (Active Comparator): MIRPE utilizing just one metallic bar
  Interventions: Procedure: MIRPE with one bar
- Two bars (Active Comparator): MIRPE utilizing two metallic bars fixed with the bridge device
  Interventions: Procedure: MIRPE with two bars

INTERVENTIONS:
Procedure: MIRPE with two bars — Minimally invasive repair of pectus excavatum utilizing two metallic bars
  Arms: Two bars
Procedure: MIRPE with one bar — Minimally invasive repair of pectus excavatum utilizing one metallic bar
  Arms: One bar

SUMMARY:
Pectus excavatum (PE) is the most common congenital deformity of the chest wall and surgical treatment using the minimally invasive technique (MIRPE) is consolidating as the choice to perform PE correction. In this technique, a temporary metal bar is placed in a retrosternal position, pushing the sternum without the need for cartilage resection. Despite the advantages obtained, it is not free from complications, with the displacement of the bar being one of the main problems. Therefore, the aim of this study is to evaluate a new bridging device for the set of two metal bars to be used in the surgical treatment of PE, verifying the clinical and surgical complications and evaluating the change in lung volumes and thoracoabdominal kinematics using optoelectronic plethysmography , preoperatively and 180 days after MIRPE; and also evaluating diaphragmatic mobility via ultrasound examination to assess the craniocaudal displacement of the left branch of the vein preoperatively and 180 days later. There will be 20 participants, who after performing a computed tomography of the chest to obtain the Haller index, clinical and laboratory tests, electrocardiogram and echocardiogram. Participants will be randomized and divided into two groups: 10 control individuals (traditional MIRPE technique used in the Service) and 10 intervention individuals (with bridge fixators developed in partnership with Traumec Tecnologia e Implantes, Brazil). The effectiveness of the fixators will be evaluated by the degree of displacement of the bars, using a mathematical formula, using a lateral chest X-ray in the immediate postoperative period (d0) and another image from the end of the period analyzed (dX), 15, 30, 90 and 180 days after the surgical procedure; evaluation of postoperative pain through the numerical pain scale; use of validated questionnaires on quality of life (physical and mental health) using two instruments, SF-36 and PEEQ. All data obtained between the two groups will be submitted to descriptive and inferential statistics.

DETAILED DESCRIPTION:
Population to be studied: 20 individuals with pectus excavatum will be selected to undergo minimally invasive repair of pectus excavatum (MIRPE). Participants will be randomized into two groups: control and intervention group. In the latter, two metal bars and the bridge model fastener will be used as proposed in this study.

The preoperative evaluation consists of anamnesis, physical examination, and laboratory tests. An electrocardiogram and echocardiogram will be performed to assess the participants' cardiac function. A computed tomography (CT) scan of the chest will also be performed to obtain the Haller index, as well as an analysis of lung volumes and thoracoabdominal kinematics and diaphragmatic mobility.

Participants will also answer the quality of life questionnaires that will be repeated postoperatively.

Participants will undergo minimally invasive repair of pectus excavatum (MIRPE) with one or two metal bars according to randomization.

In the postoperative period, the displacement of the metal bars will be evaluated through chest X-ray and pain scale evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 12 years of age;
* Pectus excavatum;
* Haller index > 3.25

Exclusion Criteria:

* Associated congenital anomalies;
* Unable to answer the quality of life questionnaires;
* Congenital heart disease;
* Chronic immunosuppression.
* Previous chest surgery or pleural drainage
* Associated coagulopathies and/or use of anticoagulant medications

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Thoracoabdominal kinematics and lung volumes | Change from baseline to 180 days
  Measurement of lung volumes in liters (L) will be obtained indirectly through optoelectronic plethysmography.
Metallic bars displacement | Change from baseline to 180 days.
  The displacement of the bars measured in millimeters (mm) in the lateral chest X-ray in the immediate postoperative (d0) and at the end of the period analyzed (dX) considering the distance between the upper point of contact of the bar with the sternum and the most posterior and superior point of the body of the sternum. The bar displacement index is calculated according to the formula: d0 - dX / d0 x 100.

SECONDARY OUTCOMES:
Diaphragmatic mobility | Pre op and 180 days
  Measurement of the craniocaudal displacement of the left branch of the portal vein in millimeters (mm) by ultrasonographic examination as a measure of diaphragmatic mobility.
Pain intensity | Change from baseline to 180 days
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Quality of life related to physical and mental health | Preoperative period and 180 days
  The Short-Form-36 Health Survey (SF-36) is a multidimensional instrument to assess health-related quality of life. It comprises two summary subscales: (1) the physical component summary features aspects of 'physical functioning', 'physical role functioning', 'bodily pain', and 'health in general' and (2) the mental component summary is based on the dimensions 'social functioning', 'emotional role functioning', 'vitality', and 'mental health'. Higher scores are indicative of better health.
Physical and psychosocial quality-of-life changes after surgical repair of pectus excavatum | Preoperative period and 180 days
  The Pectus Excavatum Evaluation Questionnaire (PEEQ) consists of 12 questions for patients which result can vary from 21 to 40; and with 13 questions for their parents which result can vary from 13 to 52 with bigger numbers representing better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L Tedde, MD, PhD, Principal Investigator — Heart Institute (InCor) FMUSP; Paulo M Pego-Fernandes, MD, PhD, Study Director — Heart Institute (InCor) FMUSP
Locations (1):
- Heart Institute (InCor) Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Carvalho RLC, Tedde ML, de Campos JRM, Hamilton NN, Guilherme GF, Sousa VM, Junior VFS, Savazzi FH, Pego-Fernandes PM. Quality of life outcomes after minimally invasive repair of pectus excavatum utilizing a new set of metallic bars and stabilizers. J Pediatr Surg. 2021 Mar;56(3):545-549. doi: 10.1016/j.jpedsurg.2020.06.036. Epub 2020 Jun 30. PMID 32711943
- [Background] Tedde ML, Togoro SY, Eisinger RS, Okumura EM, Fernandes A, Pego-Fernandes PM, Campos JRM. Back to the future: a case series of minimally invasive repair of pectus excavatum with regular instruments. J Bras Pneumol. 2019 Feb 11;45(1):e20170373. doi: 10.1590/1806-3713/e20170373. PMID 30758428
- [Background] Togoro SY, Tedde ML, Eisinger RS, Okumura EM, de Campos JRM, Pego-Fernandes PM. The Vacuum Bell device as a sternal lifter: An immediate effect even with a short time use. J Pediatr Surg. 2018 Mar;53(3):406-410. doi: 10.1016/j.jpedsurg.2017.04.016. Epub 2017 May 1. PMID 28495420
- [Background] de Campos JR, Tedde ML. Management of deep pectus excavatum (DPE). Ann Cardiothorac Surg. 2016 Sep;5(5):476-484. doi: 10.21037/acs.2016.09.02. PMID 27747181
- [Background] Tedde ML, de Campos JR, Wihlm JM, Jatene FB. The Nuss procedure made safer: an effective and simple sternal elevation manoeuvre. Eur J Cardiothorac Surg. 2012 Nov;42(5):890-1. doi: 10.1093/ejcts/ezs442. Epub 2012 Jul 24. PMID 22833539
- [Background] Tedde ML, Campos JR, Das-Neves-Pereira JC, Abrao FC, Jatene FB. The search for stability: bar displacement in three series of pectus excavatum patients treated with the Nuss technique. Clinics (Sao Paulo). 2011;66(10):1743-6. doi: 10.1590/s1807-59322011001000012. PMID 22012046